CLINICAL TRIAL: NCT05820802
Title: High Dimensional Analysis of Immune Cells Using scRNA-seq in Pediatric Patients With Allergic Reactions to Neuromuscular Blockers
Brief Title: High Dimensional Analysis of Immune Cells in Pediatric Patients
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Young-Eun Jang, Clinical Associate Professor, Seoul National University Hospital
Other Study IDs: 2208-169-1354
Record Dates: First submitted 2023-03-22; First posted 2023-04-20 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Drug Allergy; Neuromuscular Blockade
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to characterize immune cells using single-cell transcriptomic analysis in pediatric patients aged 2 to 18 years undergoing general anesthesia who are expected to receive Rocuronium, a non-depolarizing neuromuscular blocking agent, in the event of an allergic reaction.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients between the ages of 2 and 18 undergoing general anesthesia and surgery using the neuromuscular blocker, rocuronium.

Exclusion Criteria:

* Patients who have received immunomodulators, immunosuppressants, etc.
* Patients with autoimmune diseases (rheumatoid arthritis, lupus, Behcet's disease, etc.)
* Patients who regularly take, or have taken within 4 weeks, medications that may affect the immune system (oral steroids, anti-inflammatories, etc.)
* Other cases where the Principal Investigator determines that it is difficult to conduct the study.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric patients between the ages of 2 and 18 undergoing general anesthesia using the rocuronium.
Sampling Method: Non-Probability Sample
Enrollment: 294 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Transcriptomic profile analysis of the T lymphocytes by RNA sequencing | until end of surgery (usually up to 12 hours from the first dose of rocuronium)
  Blood sample from the patients when patient shows allergic reaction after administration of rocuronium

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea